CLINICAL TRIAL: NCT04411914
Title: A Phase 1B Double Blind, Placebo (PBO) Controlled, Pharmaco- Magnetic Resonance Spectroscopy (MRS) Inpatient Study of Clavulanic Acid (CLAV) 500, 750, 1000 mg Daily Repeated Administration in Early Remitted Cocaine Use Disorder Subjects
Brief Title: Pharmaco-Magnetic Resonance Spectroscopy (MRS) Study of Clavulanic Acid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); University of Pennsylvania (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 26876; U01DA048517 (NIH)
Record Dates: First submitted 2020-05-20; First posted 2020-06-02 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Clavulanic Acid; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel group inpatient study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clavulanic Acid (Experimental): Participants will receive 10 days of CLAV-- Period 1: 500 mg/day for days 1-3; Period 2: 750 mg/day for days 4-6; Period 3: 1000 mg/day for days 7-10.
  Interventions: Drug: Clavulanic Acid
- Placebo (Placebo Comparator): Participants will receive 10 days of placebo and will have a "dose" escalation at the same time as the experimental group. They will be given additional placebo pills to match the number given to the experimental group (i.e. 2 PBO capsules/day for days 1-3, 3 PBO capsules/day days 4-6 and 4 PBO capsules/day for days 7-10).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Clavulanic Acid — Drug will be given in 250mg capsules.
  Arms: Clavulanic Acid
Other: Placebo — Placebo
  Other Names: microcrystalline cellulose
  Arms: Placebo

SUMMARY:
A dose-escalation study to determine the optimum dose of Clavulanic Acid (CLAV) for effects on craving and efficacy.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel group inpatient study of clavulanic acid for 10 days in adults (18-65) seeking treatment for cocaine use disorder. For those subjects who can tolerate 500 mg/day for 3 days (or matched placebo), there will be a forced dose escalation to 750 mg/day for 3 days. Subjects who can tolerate 750 mg/day for three days will have a forced dose escalation to 1000 mg/day for 4 days until the study ends.

Thus, there are 3 Periods for each participant:

Period 1: 500 mg CLAV per day for days 1-3; Period 2: 750 mg per day for days 4-6; Period 3: 1000 mg/day for days 7-10.

Subjective, cognitive, and adverse effect assessments, blood pressure and pulse will be performed daily. Structural MRI, resting state MRI (rs-fMRI), functional MRI (fMRI) and Magnetic Resonance Spectroscopy (MRS) scans will be done at baseline and on Days 3, 6 and 10 of the study. At the time of each scan, safety of the subject to complete the scan will be re-assessed. fMRI was not done at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to verbalize understanding of consent form
2. Be male or female adult volunteers ages 18-65 inclusive.
3. Have a Diagnostic and Statistical Manual-5 (DSM-5) diagnosis of cocaine use disorder, moderate to severe in early remission
4. Have a Body Mass Index (BMI) of 17.5 to 39.9 kg/m2; and a total body weight of at least 45 kg (99 lbs.)
5. Have a history and brief physical examination that demonstrate no clinically significant contraindication for participating in the study, and/ or significant or unstable medical or psychiatric illness.

Exclusion Criteria:

1. Have a current DSM-5 substance use disorder, mild, moderate, or severe, on any drug of abuse other than nicotine, caffeine, and cocaine use disorder in early remission verified by Urine Drug Screen (UDS). Alcohol use disorder and marijuana use disorder, mild without withdrawal symptoms, will be permitted.
2. Have any previous medically adverse reaction to CLAV, Augmentin, penicillin, Ticarcillin, cephalosporin, or any beta-lactam drug.
3. Have any illness, condition, and use of medications, in the opinion of the principal investigator, sub-investigators which would preclude safe and/or successful completion of the study.
4. Report having human immunodeficiency virus (HIV) infection or test positive for HIV during screening
5. Be pregnant (females).
6. Unable to tolerate MRI scan for duration of 60 minutes for physical or psychological reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University Episcopal Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim J, John J, Langford D, Walker E, Ward S, Rawls SM. Clavulanic acid enhances glutamate transporter subtype I (GLT-1) expression and decreases reinforcing efficacy of cocaine in mice. Amino Acids. 2016 Mar;48(3):689-696. doi: 10.1007/s00726-015-2117-8. Epub 2015 Nov 5. PMID 26543027
- [Derived] Callans LS, Philogene-Khalid H, Jagannathan K, Cunningham R, Yu D, Lu X, Walters MI, Morrison MF. Clavulanic Acid Decreases Cocaine Cue Reactivity in Addiction-Related Brain Areas, a Randomized fMRI Pilot Study. Psychopharmacol Bull. 2024 Apr 4;54(2):8-14. doi: 10.64719/pb.4485. PMID 38601830

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment materials included newspapers, facebook, and word of mouth. Participants were recruited from the local community between 9/2020 and 11/2021.
Groups:
- Clavulanic Acid: 10 Participants will receive CLAV for 10 days over 3 Periods with no CLAV for Day 11.
  Period 1 CLAV 500 mg/day for 3 days dose Period 2- CLAV 750 mg/day for 3 days. Period 3 CLAV 1000mg for 4 days
  Clavulanic Acid Only Product: Drug will be given in 250mg capsules.
- Placebo: 3 participants will receive placebo and serve as a control group. They will be blinded to their condition and will have a "dose" escalation at the same time as the experimental group, and be given additional placebo pills to match the number given to the experimental group.
  Placebo: Placebo
Period: CLAV 500mg/Day for Days 1-3
Arm/Group | Clavulanic Acid | Placebo
Started | 10 | 3
Completed | 9 | 3
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: CLAV 750mg/Day for Days 4-6
Arm/Group | Clavulanic Acid | Placebo
Started | 9 (9 participants who completed Period 1 (3 days of CLAV 500mg for 3 days) had dose escalation to 750mg/d for 3 days in Period 2.) | 3
Completed | 9 | 3
Not Completed | 0 | 0
Period: CLAV 1000m/d for Days 7-10
Arm/Group | Clavulanic Acid | Placebo
Started | 9 (The same 9 participants who started the study and received 3days of CLAV 500mg/day and 3 days of CLAV 750mg/day were then dose escalated to CLAV 1000mg/day for 4 days.) | 3
Completed | 9 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clavulanic Acid: 10 participants randomized to the CLAV group
  Clavulanic Acid will be given in 250mg capsules according to the 3 Periods
- Placebo: 3 participants will receive placebo (PBO) and serve as a control group. They will have a "dose" escalation at the same time as the experimental group, and be given additional placebo pills to match the number given to the experimental group.
  Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Clavulanic Acid | Placebo | Total
Number analyzed (Participants) | 10 | 3 | 13
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54.2 [49.8 to 57.8] | 57.8 [45.3 to 60.9] | 55.6 [47.6 to 57.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 3 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 3 | 0 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 3 | 0
Handedness [Count of Participants; unit: Participants]
  left-handed | 0 | 1 | 1
  right-handed | 10 | 2 | 12
Education [Count of Participants; unit: Participants]
  Left formal education at 16 | 0 | 1 | 1
  Left formal education at 17-18 | 5 | 2 | 7
  Undergraduate or Equivalent | 4 | 0 | 4
  unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Brain Glutamate Concentration in the Anterior Cingulate Cortex (ACC) in Subjects With Cocaine Use Disorder (CUD) Treated With Escalating Doses of Clavulanate (CLAV)
Description: Brain glutamate concentration in the ACC (based on Magnetic Resonance Spectroscopy (MRS)) will be correlated with cocaine craving (measured by Cocaine Craving Questionnaire (CCQ)) in subjects receiving escalating doses of CLAV for 10 days. Measurement will be made at baseline and Day 10 of CLAV (1000 mg/day) in subjects with cocaine use disorder.
Time Frame: ACC glutamate and CCQ will be measured and correlated on Day 10 of treatment with CLAV compared with baseline.
Population: Glutamate (Glu) level (MR-Spectroscopy) in the ACC (9 scans at baseline and 9 scans at Day 10, adjusted for baseline) are correlated with CCQ results (9 baseline questionnaires and 9 day 10 questionnaires). Spearman Correlation Coefficients were calculated. Higher concentrations of ACC glutamate on day 10 correlated with decreased cocaine craving.
Measure: Number; unit: Spearman Correlation Coefficient
Units Other Than Participants: MRS Scans and CCQ
Groups:
- Clavulanic Acid Day 10: 9 participants who completed Periods 1, 2 and 3 were assessed for brain Glutamate levels in the ACC using MRS at the end of Period 3 (Day 10.)This measure was correlated with CCQ on day 10 adjusted for the baseline.
- Clavulanic Acid Baseline: Same 9 subjects underwent CCQ and MRS on Day 1 prior to receiving CLAV 500 mg.
Arm/Group | Clavulanic Acid Day 10 | Clavulanic Acid Baseline
Number analyzed (Participants) | 9 | 9
Number analyzed (MRS Scans and CCQ) | 18 | 18
Spearman Correlation Coefficient | -0.9000 | 0.3333
Statistical Analysis 1: Comparison: Clavulanic Acid Day 10; Test type: Superiority; p = 0.0009, Spearman Correlation Coefficient

2. Secondary Outcome: Changes in Resting State Network Connectivity From Baseline
Description: Craving-associated neurocircuitry (frontal-striatal-thalamic connectivity) will be examined with resting state functional Magnetic Resonance Imaging (rs-fMRI) and Cocaine Craving Questionnaire (CCQ-45). The CCQ is comprised of five 9-item sub-scales (desire to use cocaine, intention and planning to use cocaine, anticipation of positive outcome from use, anticipation of relief from withdrawal or dysphoria, and lack of control over use) measured on a scale of 1 to 7, total scores ranging from 45 to 315 with higher numbers indicating increased craving.. The rs-fMRI activity and CCQ were assessed in the 9 participants at baseline and at the end of each of 3 periods. rs-fMRI activity and CCQ were correlated using the Spearman Correlation Coefficient calculation. A negative correlation coefficient indicates an inverse relationship between the assessments; higher rs-fMRI activity correlates with lower craving.
Time Frame: Assessment was done at the end of Period 1, 2 and 3 detailed above. Data from the end of Period 3 (Day 10, 1000mg CLAV) are reported.
Population: 9 participants completed Period 1 (3 days of CLAV 500mg) Period 2 (3 days of CLAV 750mg) and then Period 3 (4 days of CLAV 1000mg). The rs-fMRI activity in the executive control network and CCQ were correlated using the Spearman Correlation calculation at the end of this course of study drug (Day 10) and are reported.
Measure: Number; unit: Spearman Correlation Coefficient
Groups:
- Rs-fMRI and CCQ on Day 10 CLAV: rs-fMRI activity of the Executive Control Network at the end of Period 3 (day 10 of CLAV (dose 1000mg/day)) adjusted for baseline was correlated with CCQ day 10. Subjects had a baseline scan on Day 1 prior to receiving CLAV 500mg. They received CLAV 500mg/day days 1-3. CLAV 750 mg/day days 4-6 and CLAV 1000 mg/day on days 7-10 and then did the CCQ and had repeat rs-fMRI on day 10.
Arm/Group | Rs-fMRI and CCQ on Day 10 CLAV
Number analyzed (Participants) | 9
Spearman Correlation Coefficient | -0.8333
Statistical Analysis 1: Comparison: Rs-fMRI and CCQ on Day 10 CLAV; Test type: Other; p = 0.0053, Spearman Correlation Coefficient; Spearman Correlation Coefficient, N=9 Prob > |r| under H0: Rho=0

3. Secondary Outcome: Craving
Description: Craving will be evaluated by Cocaine Craving Questionnaire (CCQ-45). The CCQ is comprised of five 9-item sub-scales (desire to use cocaine, intention and planning to use cocaine, anticipation of positive outcome from use, anticipation of relief from withdrawal or dysphoria, and lack of control over use) measured on a scale of 1 to 7, total scores ranging from 45 to 315 with higher numbers indicating increased craving. The results are the CCQ scores on day 10 minus the baseline scores before starting study drug.
Time Frame: CCQ-45 questionnaires were completed daily during the study. Data from day 10 adjusted for baseline score are reported.
Measure: Mean (Standard Deviation); unit: difference in score on a scale
Groups:
- Male CLAV Subjects--CCQ on Day 10: CCQ-45 scores on Day 10 in male subjects (who took CLAV 500mg/day for 3 days, then 750 mg/day for 3 days and 1000mg/day for 4 days) minus the baseline CCQ scores.
- Male PBO Subjects--CCQ Score Day 10: CCQ scores on Day 10 minus the baseline CCQ scores in male subjects who took matched PBO for 10 days.
- Female CLAV Subjects--CCQ Score Day 10: CCQ-45 scores from day 10 in female subjects (they took CLAV 500mg/3 for the first 3 days, then 750 mg/day for days for 3 days and 1000mg/day for 4 days) minus the baseline scores.
- Femaile PBO Subjects--CCQ Scores Day 10: The CCQ scores day 10 minus the baseline scores in female submects who took matched PBO for 10 days.
Arm/Group | Male CLAV Subjects--CCQ on Day 10 | Male PBO Subjects--CCQ Score Day 10 | Female CLAV Subjects--CCQ Score Day 10 | Femaile PBO Subjects--CCQ Scores Day 10
Number analyzed (Participants) | 6 | 2 | 3 | 1
difference in score on a scale | 7 (16) | -22 (10) | -15 (21) | 49 (0)

4. Secondary Outcome: Change in Brain Glutamine From Baseline
Description: Change in brain glutamine (Gln) concentration in the ACC at Day 10 compared to baseline as assessed by MRS in the ACC.
Time Frame: Brain glutamine will be analyzed at baseline (Day 1 prior to CLAV or PBO dose) and at Day 10 day (having completed Periods 1, 2 and 3 (CLAV 500mg/day for 3 days, 750 mg/day for 3 days and 1000 mg/day for 4 days).
Measure: Mean (Standard Deviation); unit: mmol/kg
Groups:
- Clavulanic Acid (CLAV) Group Baseline: Glutamine (Gln) levels measured in 9 participants by MRS in the ACC at baseline (prior to receiving any dose of CLA V)
- Clavulanic Acid Day 10: Gln levels measured in 9 participants by MRS in the ACC on Day 10 of CLAV dosing having taken CLAV 500mg for 3 days, 750 mg for 3 days and 1000 mg for 4 days.
- Placebo Group Baseline: Gln levels measured in 3 participants by MRS in the ACC at baseline (prior to receiving any dose of Placebo)
- Placebo Group Day 10: Gln levels measured in 3 participants by MRS in the ACC on Day 10 of matching Placebo.
Arm/Group | Clavulanic Acid (CLAV) Group Baseline | Clavulanic Acid Day 10 | Placebo Group Baseline | Placebo Group Day 10
Number analyzed (Participants) | 9 | 9 | 3 | 3
mmol/kg | 1.5 (1.0) | 2.1 (2.0) | 0.8 (0.3) | 0.7 (0.6)

5. Secondary Outcome: Number of Participants With Treatment-related Adverse Events (AEs)
Description: Adverse events (AES) will be defined as any clinically significant changes in vital signs, clinically significant change in Electrocardiogram (EKG) from baseline measurement, clinically significant changes in laboratory bloodwork (Complete blood count, comprehensive metabolic panel, urinalysis), or any self reported side effects compared with baseline. AEs will be collected throughout the study and reviewed by a physician. An evaluation of AE severity (mild, moderate, severe) will be evaluated by a physician based on participant self-report. AEs per subject will be listed by organ system, and the number of AEs within the subject population will be totaled.
Time Frame: 1-24 days (during and up to 2 weeks after study dosing period)
Population: see adverse events report; Blood Pressure, heart rate, EKG were not statistically different between the two groups.
Measure: Count of Participants; unit: Participants
Groups:
- Clavulanic Acid: 9 Participants will receive 500 mg of CLAV at baseline. Subjects who can tolerate 500 mg/day for 3 days (or matched placebo) will have a dose escalation to 750 mg/day for 3 days. Subjects who can tolerate 750mg/day for three days will have a dose escalation to 1000mg for 4 days.
  Clavulanic Acid Only Product: Drug will be given in 250mg capsules.
Arm/Group | Clavulanic Acid | Placebo
Number analyzed (Participants) | 10 | 3
Participants | 6 | 1

ADVERSE EVENTS:
Time Frame: 24 days
Description: 9 subjects in the CLAV group and 3 subjects in the PBO group will be assessed throughout the study for Adverse Events (AE).
  Subjects in the CLAV group are treated in 3 periods: CLAV 500 mg for 3 days, 750mg for the next 3 days and then 1000mg for the last 4 days to complete the 10 days of the study. AEs were reported by period/dose though the same person may have had several AE or the same AE at different doses.
Groups:
- Clavulanic Acid Treatment Period 1-500mg/Day: 10 Participants will be treated with CLAV (500mg/day for 3 days)
- CLavulanic Acid Treatment Period 2-750mg.Day: 9 Participants who completed Period 1 treated with CLAV (750mg/day for 3 days)
- Clavulanic Acid Treatment Period 3--1000mg/Day: 9 Participants who completed Period 1 treated with CLAV (1000mg/day for 3 days)
- Placebo: 3 participants received matched placebo. They will be given additional placebo capsules to match the number given to the CLAV group.
Arm/Group | Clavulanic Acid Treatment Period 1-500mg/Day | CLavulanic Acid Treatment Period 2-750mg.Day | Clavulanic Acid Treatment Period 3--1000mg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 6/10 | 5/9 | 2/9 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clavulanic Acid Treatment Period 1-500mg/Day (N=10) | CLavulanic Acid Treatment Period 2-750mg.Day (N=9) | Clavulanic Acid Treatment Period 3--1000mg/Day (N=9) | Placebo (N=3)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1
flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
loose stool (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (2)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated Liver Function Tests (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Drug induced hepatitis, asymptomatic, resolved in 2 weeks, discontinued from study
High blood pressure (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Swollen feet (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Lightheaded (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Priapism (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT04411914/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT04411914/ICF_001.pdf